CLINICAL TRIAL: NCT02236611
Title: A Randomized, Parallel-group, Open-label Study to Evaluate the Efficacy and Safety of Umeclidinium (UMEC) 62.5 mcg Compared With Glycopyrronium 44 mcg in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A 12-week Study to Evaluate the Efficacy and Safety of Umeclidinium 62.5 Microgram (mcg) Compared With Glycopyrronium 44 mcg in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201315
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; inhaler ease of use; glycopyrronium; umeclidinium; novel dry powder inhaler; long-acting muscarinic antagonist; inhaler errors
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umeclidinium 62.5 mcg (Experimental): Randomized subjects will receive umeclidinium inhalation powder 62.5 mcg, once daily over a period of 12 weeks via a nDPI. Subjects will be instructed to take one dose each morning.
  Interventions: Drug: Umeclidinium
- Glycopyrronium 44 mcg (Experimental): Randomized subjects will receive glycopyrronium 44 mcg, once daily over a period of 12 weeks via a BREEZHALER inhaler. Subjects will be instructed to take one dose each morning.
  Interventions: Drug: Glycopyrronium

INTERVENTIONS:
Drug: Umeclidinium — Umeclidinium 62.5 mcg will be available as dry inhalation powder to be taken using a nDPI
  Arms: Umeclidinium 62.5 mcg
Drug: Glycopyrronium — Glycopyrronium bromide will be available as inhalation capsules, 44 mcg per capsule, taken using BREEZHALER inhalers
  Arms: Glycopyrronium 44 mcg

SUMMARY:
This is a 12-week, multicentre, randomized, open-label, 2-arm, parallel-group study designed to compare the efficacy and safety of umeclidinium inhalation powder (62.5 mcg once daily [QD]) administered via a novel Dry Powder Inhaler (nDPI) with glycopyrronium (44 mcg QD) administered via a Breezhaler® inhaler in subjects with COPD over 12 weeks of treatment. At the end of the run-in period, eligible subjects will be randomized in a 1:1 ratio to receive umeclidinium 62.5 mcg administered via nDPI or glycopyrronium 44 mcg administered via BREEZHALER inhaler. There will be up to 8 clinic visits conducted on an outpatient basis at Pre-Screening (Visit 0), Screening (Visit 1), Randomization at Day 1 (Visit 2), and after Randomization at Day 2 (Visit 3), Day 28 (Visit 4), Day 56 (Visit 5), Day 84 (Visit 6) and Day 85 (Visit 7). The total duration of subject participation in the study will be approximately 15 weeks. The primary endpoint of the study is clinic visit trough FEV1 (forced expiratory volume in one second) on treatment Day 85. All subjects will have spirometry performed at clinic Visits 1 though 7. Trough spirometry will be obtained 23 and 24 hours after the previous day's dose of open-label study medication at Visits 3 to 7.

BREEZHALER is a registered trademark of Novartis AG.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: outpatient
* Informed Consent: a signed and dated written informed consent prior to study participation
* Age: subjects 40 years of age or older at Visit 1.
* Gender: male and female subjects are eligible to participate in the study. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile. Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, eg, age appropriate, > 45 years, in the absence of hormone replacement therapy OR child bearing potential, has a negative pregnancy test at screening, and agrees to one of the acceptable contraceptive methods used consistently and correctly i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact.
* Diagnosis: an established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society (ERS)
* Smoking history: current or former cigarette smokers with a history of cigarette smoking of >= 10 pack-years [number of pack years = (number of cigarettes per day / 20) x number of years smoked (eg. 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years both equal 10 pack-years)]. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack-year history
* Severity of Disease: A pre and post-albuterol/salbutamol forced expiratory volume in one second/ forced vital capacity (FEV1/FVC ratio of <0.70 and a post-albuterol/salbutamol FEV1 of >=30% and =<70% of predicted normal values at Visit 1. Predicted values will be based upon the ERS Global Lung Function Initiative
* Dyspnea: A score of >=2 on the modified medical research council dyspnea scale (mMRC) at Visit 1

Exclusion Criteria:

* Pregnancy: women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: a current diagnosis of asthma.
* Other respiratory disorders: known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease.
* Other diseases/abnormalities: any subject who is considered unlikely to survive the duration of the study period or has any rapidly progressing disease or immediate life-threatening illness (e.g. cancer). In addition, any subject who has any condition (e.g. neurological condition) that is likely to affect respiratory function should not be included in the study.
* Severe hepatic impairment: patients with severe hepatic impairment (Child-Pugh class C) should be excluded unless, in the opinion of the investigator, the benefit is likely to outweigh the risk.
* Severe renal impairment: patients with severe renal impairment (e.g., end-stage renal disease requiring dialysis) should be excluded, unless in the opinion of the investigator, the benefit is likely to outweigh the risk.
* Unstable or life threatening cardiac disease: long-acting muscarinic antagonists (LAMA) should be used with caution in subjects with severe cardiovascular disease. In the opinion of the investigator, use should only be considered if the benefit is likely to outweigh the risk in conditions such as: Myocardial infarction or unstable angina in the last 6 months, Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months, New York Heart Association (NYHA) Class IV heart failure
* Contraindications: Any history of allergy or hypersensitivity to any anticholinergic/ muscarinic receptor antagonist, sympathomimetic, lactose/milk protein or magnesium stearate.
* Antimuscarinic effects: Subjects with medical conditions such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy, or bladder neck obstruction should only be included if, in the opinion of the study physician, the benefit outweighs the risk.
* Hospitalization: hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung resection: lung volume reduction surgery within the 12 months prior to Visit 1.
* 12-Lead electrocardiogram (ECG): Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. The Investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. Subjects with the following abnormalities are excluded from participation in the study: Atrial fibrillation with rapid ventricular rate >120 beats per minute; sustained or nonsustained ventricular tachycardia; second degree heart block Mobitz type II or third degree heart block (unless pacemaker or defibrillator had been inserted)
* Medication prior to spirometry: unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Medications prior to screening: use of the following medications according to the following defined time intervals prior to Visit 1: depot corticosteroids 12 weeks, systemic, oral or parenteral corticosteroids 6 weeks, antibiotics (for lower respiratory tract infection) 6 weeks, inhaled long acting beta2 agonists/ inhaled corticosteroid (LABA/ICS) combination products if LABA/ICS therapy is discontinued completely 30 days; LABA/ICS combination products only If discontinuing ICS/ LABA therapy and switching to ICS monotherapy 48 hours for the salmeterol or formoterol component 14 days for the vilanterol component (note: the dose of ICS must be a dose of fluticasone propionate (FP) or equivalent but not to exceed 1000 mcg/day), use of ICS at a dose >1000 microgram (mcg)/day of FP or equivalent 30 days (note: use of ICS is permitted provided the dose does not exceed 1000 mcg of FP or equivalent; ICS use not to be initiated or discontinued within 30 days prior to Visit 1, except for subjects on LABA/ICS therapy who may discontinue the ICS/LABA product as indicated in the table above and switch to ICS monotherapy); initiation or discontinuation of ICS use 30 days (note: use of ICS is permitted provided the dose does not exceed 1000 mcg of FP or equivalent; ICS use not to be initiated or discontinued within 30 days prior to Visit 1, except for subjects on LABA/ICS therapy who may discontinue the ICS/LABA product as indicated in the table above and switch to ICS monotherapy); phosphodiesterase 4 (PDE4) Inhibitor (roflumilast) 14 days; LABA: salmeterol and formoterol 48 hours; olodaterol, indacaterol, and vilanterol 14 days; LAMA: tiotropium, aclidinium, glycopyrronium, umeclidinium 7 days; LAMA/LABA combination products if LAMA/LABA therapy is discontinued completely then apply whichever mono component has the longest washout; theophyllines 48 hours; Oral beta2-agonists: long-acting 48 hours, short-acting 12 hours; inhaled short acting beta2-agonists 4 hours (note: use of study provided albuterol/salbutamol is permitted during the study, except in the 4-hour period prior to spirometry testing); inhaled short-acting anticholinergics 4 hours; inhaled short-acting anticholinergic/short-acting beta2-agonist combination products 4 hours; any other investigational medication 30 days or within 5 drug half-lives (whichever is longer).
* Oxygen: use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e. =<12 hours per day) is not exclusionary.
* Nebulized therapy: regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g. albuterol/salbutamol) via nebulized therapy.
* Pulmonary rehabilitation program: participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or alcohol abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with investigator site: is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Inability to read: in the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Actual)
Dates: Start 2014-09-26 (Actual); Primary Completion 2015-06-02 (Actual); Study Completion 2015-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (72):
- Argentina (6):
  - GSK Investigational Site, Paraná, Buenos Aires
  - GSK Investigational Site, Concepción del Uruguay, Entre Ríos Province
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Chile (5):
  - GSK Investigational Site, Talca, Maule Region
  - GSK Investigational Site, Concepción, Región Del Biobio
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Czechia (7):
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Lovosice
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Rudna U Prahy
  - GSK Investigational Site, Třebíč
  - GSK Investigational Site, Varnsdorf
- Germany (11):
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Brinkum/Stuhr, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
- Hungary (6):
  - GSK Investigational Site, Balassagyarmat
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Kapuvár
  - GSK Investigational Site, Nagykanizsa
  - GSK Investigational Site, Törökbálint
- Norway (7):
  - GSK Investigational Site, Ålesund
  - GSK Investigational Site, Hakadal
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Hønefoss
  - GSK Investigational Site, Kolbjørnsvik
  - GSK Investigational Site, Kongsvinger
  - GSK Investigational Site, Løvenstad
- Romania (7):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- Russia (16):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Chita
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petesburg
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Yekaterinburg
- Spain (5):
  - GSK Investigational Site, Laredo, Cantabria
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Fuenlabrada / Madrid
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Peralada( Girona)
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Shah D, Driessen M, Risebrough N, Baker T, Naya I, Briggs A, Ismaila AS. Cost-effectiveness of umeclidinium compared with tiotropium and glycopyrronium as monotherapy for chronic obstructive pulmonary disease: a UK perspective. Cost Eff Resour Alloc. 2018 May 10;16:17. doi: 10.1186/s12962-018-0101-3. eCollection 2018. PMID 29773969
- [Derived] Rheault T, Khindri S, Vahdati-Bolouri M, Church A, Fahy WA. A randomised, open-label study of umeclidinium versus glycopyrronium in patients with COPD. ERJ Open Res. 2016 Apr 27;2(2):00101-2015. doi: 10.1183/23120541.00101-2015. eCollection 2016 Apr. PMID 27730198
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 201315 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201315 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201315 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201315 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201315 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201315 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201315 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1290 par. were screened; 1037 par. were randomized and 1034 were in the ITT population which comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period. Two par. were randomized in error and one par. was randomized, but did not take any study medication.
Pre-assignment Details: Participants, with clinical history of chronic obstructive pulmonary disease, who meet the eligibility criteria at screening were enrolled in a 7 to 14 day run-in period. Participant meeting continuation criteria, during run-in period, were randomized (1:1) to receive umeclidinium or glycopyrronium.
Groups:
- UMEC 62.5 mcg QD: Participants received Umeclidinium (UMEC) inhalation powder 62.5 microgram (mcg) once-daily (QD) in morning via a novel dry powder inhaler (nDPI) for 12 weeks. Participants also received albuterol/salbutamol via metered-dose-inhaler (MDI) or nebules as needed throughout the study.
- GLYCO 44 mcg QD: Participants received glycopyrronium bromide (GLYCO) inhalation capsules 44 mcg QD in morning via an alternative dry powder inhaler (DPI) for 12 weeks. Participants also received albuterol/salbutamol via MDI or nebules as needed throughout the study.
Period: Overall Study
Arm/Group | UMEC 62.5 mcg QD | GLYCO 44 mcg QD
Started | 516 | 518
Completed | 490 | 484
Not Completed | 26 | 34
Not completed — Adverse Event | 10 | 16
Not completed — Lack of Efficacy | 4 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol deviation | 3 | 5
Not completed — Withdrew consent | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UMEC 62.5 mcg QD | GLYCO 44 mcg QD | Total
Number analyzed (Participants) | 516 | 518 | 1034
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.35) | 64.0 (8.26) | 64.1 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 168 | 329
  Male | 355 | 350 | 705
Race/Ethnicity, Customized [Number; unit: Participants]
  Central/South Asian Heritage (HRTG) | 3 | 0 | 3
  Japanese/East Asian Heritage/South East Asian HRTG | 0 | 1 | 1
  White | 513 | 517 | 1030

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 on Day 85
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Day 85 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Day 84 (Week 12). Trough FEV1 measurements were taken electronically by spirometry on Days 2, 28, 56, 84 and 85. Baseline trough FEV1 is the mean of the two assessments made -30 and -5 minutes (min) pre-dose on Day 1. Change from baseline was calculated as the trough FEV1 value on Day 85 minus the BL value. Analysis performed using a repeated measures model with covariates of treatment, baseline FEV1, centre group, 24 hour subset flag, Day, Day by baseline and Day by treatment interactions. The least squares mean changes are presented here.
Time Frame: Baseline (BL) and Day 85
Population: Per Protocol(PP) Population(pop): Participants(par) in the Intent-To-Treat pop who did not have a full protocol deviation considered to impact efficacy. Par represent those with data available at time point presented; however, all par. in the PP pop. without missing covariate information and >=1 post BL measurement are included in analysis
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | UMEC 62.5 mcg QD | GLYCO 44 mcg QD
Number analyzed (Participants) | 431 | 425
Liter | 0.123 (0.0105) | 0.099 (0.0105)
Statistical Analysis 1: Comparison: UMEC 62.5 mcg QD vs GLYCO 44 mcg QD; Test type: Non-Inferiority or Equivalence — Alternate hypothesis: the difference between the trt means (umeclidinium minus glycopyrronium) would be > -50 milliliters (mL). If the lower CI (2.5% 1-sided significance level) of the statistical test should fall above -50 mL, then umeclidinium may be deemed statistically non-inferior to glycopyrronium. If the lower CI (2.5% 1-sided significance) of the statistical testing exceeded 0 then, umeclidinium may be deemed statistically superior to glycopyrronium; p = 0.100, Mixed Models Analysis; Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.005 to 0.054]

ADVERSE EVENTS:
Time Frame: On-treatment(trt) non-serious adverse events(AEs) and serious AEs are events occurring while par were on trt or events with an onset during follow-up period(up to 13 weeks).
Description: On-treatment SAEs and non-serious AEs were reported for the Intent-To Treat Population comprised all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Arm/Group | UMEC 62.5 mcg QD | GLYCO 44 mcg QD
Serious Adverse Events (participants affected / at risk) | 17/516 | 15/518
Other Adverse Events (participants affected / at risk) | 77/516 | 80/518
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 62.5 mcg QD (N=516) | GLYCO 44 mcg QD (N=518)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 62.5 mcg QD (N=516) | GLYCO 44 mcg QD (N=518)
Nasopharyngitis (Infections and infestations) | 42 | 39
Headache (Nervous system disorders) | 42 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.